CLINICAL TRIAL: NCT02873689
Title: A Phase 3 Double-blind Study to Evaluate the Efficacy and Safety of Dexlansoprazole (30 mg QD) Compared to Placebo on Heartburn Relief in Subjects With Symptomatic Nonerosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Efficacy and Safety of Dexlansoprazole on Heartburn Relief in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-390MR_302; U1111-1171-1002 (Registry Identifier: WHO)
Record Dates: First submitted 2016-08-17; First posted 2016-08-19 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Heartburn; Gastroesophageal Reflux Disease
Keywords: Drug therapy
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, delayed-release capsule, orally, once daily for up to 4 weeks.
  Interventions: Drug: Dexlansoprazole
- Placebo (Experimental): Dexlansoprazole placebo-matching capsules, orally, once daily for up to 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole delayed-release capsule
  Arms: Dexlansoprazole 30 mg
Drug: Placebo — Dexlansoprazole placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of dexlansoprazole compared to placebo in relief of daytime and nighttime heartburn over 4 weeks in Chinese participants with symptomatic non-erosive Gastroesophageal Reflux Disease (GERD).

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to treat heartburn in people who have non-erosive gastroesophageal reflux disease (GERD). This study will look at heartburn relief in people who take dexlansoprazole.

The study will enroll approximately 200 participants. Participants will be randomly assigned to one of the two treatment groups with 1:1 ratio -which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Dexlansoprazole 30 mg
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient.

All participants will be asked to take one capsule at the same time each day throughout the study, and will be asked to record any time they have heartburn symptoms in a diary.

This multi-center trial will be conducted in China. The overall time to participate in this study is up to 7 weeks. Participants will make 4 visits to the clinic, and will be contacted by telephone 5 to 10 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants identifying their main symptom as a burning feeling in the mid-epigastric area and/or chest area (that is, heartburn).
2. Must have a history of symptomatic GERD for 6 months or longer prior to Screening with GERD symptoms that were responsive to acid-suppressive therapy.
3. Must have episodes of heartburn for 4 or more days during the 7 days prior to Day -1 as recorded in the eDiary.

Exclusion Criteria:

1. Has a history of cancer (except basal cell carcinoma of the skin), that has not been in remission for at least 5 years prior to Screening.
2. Has a known history of Barrett's esophagus with dysplastic changes or any changes suspicious Barrett's seen during screening endoscopy.
3. Participant developed acute upper gastrointestinal bleeding, gastric ulcer (a mucosal defect with white coating) or duodenal ulcer (a mucosal defect with white coating), within 30 days before the start of the Screening Visit (with the possible inclusion of those with gastric or duodenal erosion). The participant requires chronic use (greater than [>] 12 doses per month) of nonsteroidal anti-inflammatory drugs (NSAIDs) including cyclooxygenase-2 (COX-2) NSAIDs within 30 days prior to the Screening Period and throughout the study.
4. Has comorbidities that could affect the esophagus (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal strictures); a history of radiotherapy or cryotherapy of the esophagus; and a history of corrosive or physiochemical injury (with the possible inclusion in the study of those with Schatzki's ring).
5. Has a history of surgical procedures that may affect the esophagus (example, fundoplication and mechanical dilatation for esophageal strictures) or a history of gastric or duodenal surgery other than endoscopic removal of benign polyps.
6. Has erosive esophagitis (EE) as shown by endoscopy, during the Screening Period.
7. Is known to have acquired immunodeficiency syndrome (AIDS) or hepatitis, including hepatitis virus carriers: (that is, hepatitis B surface antigen HBs-antigen (HBsAg) positive or hepatitis C virus (HCV)-antibody positive).
8. Has current or historical evidence of Zollinger-Ellison syndrome or a history of gastric acid hypersecretion.
9. Is scheduled for surgery that requires hospitalization or requires surgical treatment during his/her participation in the study.
10. Has donated or lost >300 milliliter (mL) blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
11. Has a history of alcohol abuse (defined as any illicit drug use), or drug addiction in the 12 months prior to Screening.
12. Participant with positive serology result of Helicobacter pylori (H. pylori) that needs eradication therapy during the study participation period as anticipated by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (25):
- China (25):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chong Qing
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Affilicated Hospital of Guilin Medical University, Haikou, Gui Lin
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Taihe Hospital, Shiyan, Hubei
  - Central Hospital of Wuhan, Wuhan, Hubei
  - Puai Hospital Of Wuhan City, Wuhan, Hubei
  - The Third Hospital of Changsha, Changsha, Hunan
  - Zhongda Hospital Southeast, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Wuxi, Jiangsu
  - Wuxi people's hospital, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Liaocheng Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital,Sichuan University, Chengdu, Si Chuang
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- See also: Dexlansoprazole Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in China from 27 December 2016 to 19 April 2018.
Pre-assignment Details: Participants with diagnosis of symptomatic nonerosive gastroesophageal reflux disease (GERD) were enrolled in 1 of the 2 treatment groups: to receive dexlansoprazole 30 mg or placebo.
Groups:
- Placebo: Dexlansoprazole placebo-matching capsule, orally, once daily for up to 4 weeks.
- Dexlansoprazole 30 mg: Dexlansoprazole 30 mg, capsule, orally, once daily for up to 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Dexlansoprazole 30 mg
Started | 109 | 108
Treated | 108 | 107
Completed | 102 | 103
Not Completed | 7 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Randomized but not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexlansoprazole 30 mg | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.73) | 43.6 (13.24) | 44.3 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 60 | 125
  Male | 43 | 47 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 108 | 107 | 215
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 108 | 107 | 215
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.935 (3.4352) | 23.701 (3.5768) | 23.819 (3.5002)
Helicobacter pylori status [Count of Participants; unit: Participants]
  Positive | 41 | 40 | 81
  Negative | 67 | 67 | 134
Number of days with day and nighttime heartburn between study days -8 to -2 [Mean (Standard Deviation); unit: days] | 6.1 (1.27) | 6.1 (1.06) | 6.1 (1.17)
Number of days with nighttime heartburn between study days -8 to -2 [Mean (Standard Deviation); unit: days] — Population: The safety analysis set where participants for nighttime heartburn at baseline were available.
  days
    number analyzed (Participants) | 108 | 106 | 214
    (all) | 5.2 (1.83) | 5.3 (1.60) | 5.2 (1.71)
Number of days with daytime heartburn between study days -8 to -2 [Mean (Standard Deviation); unit: days] — Population: The safety analysis set where participants for daytime heartburn at baseline were available.
  days
    number analyzed (Participants) | 105 | 107 | 212
    (all) | 5.6 (1.45) | 5.3 (1.61) | 5.5 (1.54)
Severity of GERD symptoms: heartburn [Count of Participants; unit: Participants]
  None | 0 | 0 | 0
  Mild | 29 | 33 | 62
  Moderate | 56 | 55 | 111
  Severe | 22 | 17 | 39
  Very Severe | 1 | 2 | 3
Severity of GERD symptoms: acid regurgitation [Count of Participants; unit: Participants]
  None | 27 | 33 | 60
  Mild | 42 | 43 | 85
  Moderate | 27 | 24 | 51
  Severe | 12 | 6 | 18
  Very Severe | 0 | 1 | 1
Severity of GERD symptoms: dysphagia [Count of Participants; unit: Participants]
  None | 101 | 103 | 204
  Mild | 7 | 4 | 11
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0
  Very Severe | 0 | 0 | 0
Severity of GERD symptoms: belching [Count of Participants; unit: Participants]
  None | 59 | 62 | 121
  Mild | 38 | 37 | 75
  Moderate | 9 | 6 | 15
  Severe | 2 | 2 | 4
  Very Severe | 0 | 0 | 0
Severity of GERD symptoms: epigastric pain [Count of Participants; unit: Participants]
  None | 95 | 88 | 183
  Mild | 11 | 16 | 27
  Moderate | 2 | 2 | 4
  Severe | 0 | 1 | 1
  Very Severe | 0 | 0 | 0
Number of days with rescue medication use [Mean (Standard Deviation); unit: days] | 1.7 (2.68) | 0.9 (1.48) | 1.3 (2.19)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days With Neither Daytime Nor Nighttime Heartburn During Treatment
Description: The percentage of days with neither daytime nor nighttime heartburn was equal to (=) (the days that were heartburn-free during the treatment period) / (total number of days for which either a daytime or nighttime result was marked during treatment period)*100 percent (%).
Time Frame: Up to Week 4
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had post-baseline (post Day-1) data for the appropriate efficacy variables.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | Dexlansoprazole 30 mg
Number analyzed (Participants) | 108 | 107
percentage of days | 32.67 [0.0 to 100.0] | 51.72 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 30 mg; Test type: Superiority; p = 0.057, Wilcoxon rank-sum test

2. Secondary Outcome: Percentage of Days Without Nighttime Heartburn During Treatment
Description: The percentage of days without nighttime heartburn was = (the days that were heartburn-free during the treatment period) / (total number of days for which nighttime result was marked during treatment period)*100%.
Time Frame: Up to Week 4
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | Dexlansoprazole 30 mg
Number analyzed (Participants) | 108 | 107
percentage of days | 54.67 [0.0 to 100.0] | 67.86 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 30 mg; Test type: Superiority; p = 0.268, Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blind study drug (approximately Week 8).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Dexlansoprazole 30 mg
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/108 | 1/107
Other Adverse Events (participants affected / at risk) | 15/108 | 9/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Dexlansoprazole 30 mg (N=107)
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Dexlansoprazole 30 mg (N=107)
Upper respiratory tract infection (Infections and infestations) | 8 | 5
Nasopharyngitis (Infections and infestations) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT02873689/SAP_000.pdf
  • Study Protocol (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02873689/Prot_001.pdf